CLINICAL TRIAL: NCT05232110
Title: Compassionate Use of Pozelimab
Status: Approved for marketing | Type: Expanded Access
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: R3918-Pozelimab
Record Dates: First submitted 2022-01-28; First posted 2022-02-09 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: CD55-deficient Protein-losing Enteropathy
Keywords: Complement Hyperactivation, Angiopathic thrombosis, Protein-Losing Enteropathy (CHAPLE disease)
MeSH Terms: conditions — Protein-Losing Enteropathies

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Pozelimab
  Other Names: REGN3918

SUMMARY:
Provide compassionate use of pozelimab

DETAILED DESCRIPTION:
Compassionate Use requests are only being considered in response to Individual Patient Investigational New Drug (IND) applications.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult